CLINICAL TRIAL: NCT01984658
Title: A Prospective, Open Phase I Study to Investigate the Tolerability and Efficacy of Administering ALECSAT to Pancreas Cancer Patients
Brief Title: A Prospective, Open Phase I Study to Investigate the Tolerability and Efficacy of ALECSAT to Pancreas Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytoVac A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-004; 2013-001907-35 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alecsat (Experimental): The ALECSAT CBMP will be administered as single dose at week 4, 7 and week 10 which is considered an appropriate time for ALECSAT CBMP to strengthen the immune system and thus have the ability to kill tumour cells. It is the aim that the patients will receive three doses during the study period however, if the patient wish and it is recommended by the investigator, patients may receive more than three doses, continuing until progression or as judged by the Investigator. Continued treatment after the 24 week study period is only possible under the condition that no safety issues have been discovered. The interval between injections for continued treatment will be decided based on e.g. tumour response and clinical examinations.
  Interventions: Biological: Alecsat

INTERVENTIONS:
Biological: Alecsat — The ALECSAT CBMP will be administered as single dose at week 4, 7 and week 10 which is considered an appropriate time for ALECSAT CBMP to strengthen the immune system and thus have the ability to kill tumour cells. It is the aim that the patients will receive three doses during the study period however, if the patient wish and it is recommended by the investigator, patients may receive more than three doses, continuing until progression or as judged by the Investigator. Continued treatment after the 24 week study period is only possible under the condition that no safety issues have been discovered. The interval between injections for continued treatment will be decided based on e.g. tumour response and clinical examinations.

SUMMARY:
This study is a prospective open phase-I study to investigate the safety and tolerability for administration of repeated doses of ALECSAT.

Each patient will be followed up to 24 weeks from the initial blood donation to the last visit. However, the actual treatment starts on day 26, when the first single dose of ALECSAT is administered. The following administrations are given with 3 weeks intervals, i.e. at week 7 and 10. The patients are attending Kirurgisk afdeling K, Bispebjerg Hospital, and are followed by close examinations during the study period and at regular visits after completing the study as advised by the patient's responsible physician.

DETAILED DESCRIPTION:
This study is a prospective open phase-I study to investigate the safety and tolerability for administration of repeated doses of ALECSAT.

Each patient will be followed up to 24 weeks from the initial blood donation to the last visit. However, the actual treatment starts on day 26, when the first single dose of ALECSAT is administered. The following administrations are given with 3 weeks intervals, i.e. at week 7 and 10. The patients are attending Kirurgisk afdeling K, Bispebjerg Hospital, and are followed by close examinations during the study period and at regular visits after completing the study as advised by the patient's responsible physician.

The selected group of patients suffers from locally advanced pancreatic cancer and have been treated with first line treatment regimens (e.g. surgery, radiotherapy, and/or Folfirinox) and are followed at Kirurgisk afdeling K, Bispebjerg Hospital. The subjects will be recruited consecutively and included to the study if they fulfil the inclusion criteria and do not meet any of the exclusion criteria. Potential candidates will receive oral information by the Investigator subsequent to the written patient information. The potential candidate must have the opportunity to consider the given information and to further ask the Investigator questions before finally deciding to participate. When the patient decides to take part in the study he/she will be required to sign the declaration of consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from locally advanced pancreatic cancer and have started treatment with Folfirinox but must stop because of side effects or who declined the Folfirinox treatment.
* Minimum age of 18 years old and be capable of understanding the information and giving informed consent,
* Minimum height of 155 cm,
* Expected survival time (life expectancy) of over 6 months,
* Adequate performance status £ 2 (see below*),

Exclusion Criteria:

* Evident signs of distant metastasis at baseline
* Positive tests for anti-HIV-1/2; HBsAg, anti-HBc, Anti-HCV or being positive in a Treponema Pallidum test (syphilis),
* Patient´s which have visit an area where there is an outbreak of West Nile virus or Dengue virus within 28 days prior to donation should be excluded, unless the patient has been tested negative,
* Concurrent illness, e.g. uncontrolled epilepsy, cardiovascular-, cerebrovascular-, and/or respiratory disease which can worsen or cause complications in connection with blood donation,
* Clinically significant autoimmune disorders or conditions of immune suppression,
* Haemoglobin count ≤ 7.5 mmol/l (men & women),
* Lymphocytes below 0.3 x 109/l,
* Clinically abnormal Erythrocyte Volume Fraction (EVF),
* Body weight below 40 kg (men) and 50 kg (women),
* Pregnant or breast feeding women. Fertile women can only be included with a negative pregnancy test at screening and must use contraceptives during the study,
* Patients with uncontrolled serious bacterial, viral, fungal or parasitic infection,
* Blood transfusions within 48 hours prior to donation of blood for ALECSAT production,
* Any medical condition that will render participation in the study risky or, according to the investigator will make the assessment of the study endpoints difficult,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 24 weeks
  Investigation of the safety and tolerability of administrating repeated doses of ALECSAT will be measured by recording the presence of adverse events/serious adverse events during the study period, and by following clinically significant changes in blood parameters, performance status and quality of life questionnaire at specific time points and compare with the individual patients status at baseline

SECONDARY OUTCOMES:
Efficacy; Tumor change | Up to 24 weeks
  Assessment of any change in tumour involvement are followed by CT (according to the RECIST 11 protocol) at specific time points and will be compared with the individual patients status at baseline

OTHER OUTCOMES:
Efficacy; Lab parameters | Up to 24 weeks
  Changes in pancreatic cancer marker CA19-9, change in Haemoglobin, Lymphocytes and their subpopulations, Leucocytes, ASAT, ALAT, Amylase, Bilirubin, Glucose, LDH, Sodium and Potassium that may show trends of clinical effect at specific time points and will be compared with the individual patients status at baseline,
Safety & efficacy; Quality of life | Up to 24 weeks
  Changes in the patients quality of life and performance status are measured at specific time points and will be compared with the individual patients status at baseline,

CONTACTS AND LOCATIONS:
Overall Officials: Lars T. Sørensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Kirurgisk afdeling K, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
phase 1 safety study